CLINICAL TRIAL: NCT06927401
Title: Evaluate the Detection of Retained Gastric Contents and Assess Safety Using the Flower Capsule Endoscopy in Healthy Individuals and GLP-1 Receptor Agonist Users
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Endiatx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ETX-IND-01
Record Dates: First submitted 2025-04-02; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Endoscopy, Digestive System; GLP1-R-related Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The anesthesia team will be blinded to the Flower findings, and the EGD will proceed according to the standard clinical care to determine the appropriate anesthesia type and airway management approach. After 2 hours, a sedated EGD will be performed. A blinded gastroenterologist will review the images to determine the presence or absence of gastric content. Patient tolerance and Adverse Events will be documented. To minimize bias, the gastroenterologist interpreting the EGD images will be blinded to the finding of the Flower capsule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1-Fasting throughout Evaluation period (Experimental): In Group 1, participants will fast for 8 hours for food and 2 hours for clear fluids before undergoing a sedated EGD to confirm an empty stomach, serving as the ground truth. The procedure time, patient tolerance, presence or absence of gastric contents, and any adverse events (AEs) will be documented. After the fasting period and EGD, participants will consume 100 mL of water containing 400 mg of simethicone upon regaining full alertness. If necessary, they may engage in light walking and avoid prolonged sitting. After a 10-minute waiting period, they will consume an additional 100 mL of water and attempt to empty their bladder. Another 10-minute waiting period will follow, during which participants will continue drinking until they feel full, with a typical intake ranging from 500 to 1400 mL of water. If gastric distention is insufficient, additional water ingestion will be required, with the total volume documented. A blinded gastroenterologist, unaware of the participant's fasting
  Interventions: Device: Flower
- Group 2- Fasting till 8 hours and fed during Evaluation period (Experimental): In Group 2, participants will follow the same fasting protocol as Group 1, with 8 hours of fasting for food and 2 hours for clear fluids, followed by a sedated EGD to confirm an empty stomach. The procedure time, patient tolerance, presence or absence of gastric contents, and AEs will be documented. After the fasting period and EGD, participants will consume 1.5 mL/kg of a standardized food mixture -representing the minimum volume associated with high aspiration risk-once participants have fully regained alertness. Participants will consume 100 mL of water with 400 mg of simethicone. As in Group 1, if necessary, they may engage in light walking and avoid prolonged sitting. After a 10-minute waiting period, they will consume an additional 100 mL of water and attempt to empty their bladder. Another 10-minute waiting period will follow, during which they will continue drinking until they feel full, with a typical intake ranging from 500 to 1000 mL of water.
  Interventions: Device: Flower
- GLP 1 Participants (Experimental): Participants will continue taking their GLP-1 medication up to the day of the procedure. The participant will arrive at the hospital in the morning after following a 8 hour food fast and 2 hours for clear fluids. Following the fasting period, they will consume 100 mL of water containing 400 mg of simethicone. If necessary, participants should engage in light walking and avoid prolonged sitting. A 10-minute waiting period will then ensue, after which they will consume an additional 100 mL of water and attempt to empty their bladder. Another 10-minute waiting period will follow, during which participants will be instructed to drink at least 500 mL of water, continuing until a sensation of fullness is reached, with a typical total intake ranging from 500 mL to 1400 mL. If gastric distention is insufficient, additional water ingestion will be required, with the total volume documented. The Flower capsule will then be administered.
  Interventions: Device: Flower

INTERVENTIONS:
Device: Flower — Flower is a single-use capsule endoscope designed for timely visualization of the human stomach. The patient drinks water to fill the stomach before swallowing the Flower capsule, which transmits wireless video, through an external dongle placed near the patient's abdomen, to a physician's computer or smartphone. Flower is weighted to orientationally bias the capsule upward, meaning that with a few simple position adjustments a complete viewing of the stomach can be achieved approximately 10 minutes.
  The procedure requires no sedation or equipment other than the Flower System (capsule and dongle). As a simple means of screening, Flower functions equivalent to comparable technologies, but offers advantages of being less invasive and burdensome. Flower has fewer potentially adverse consequences than traditional endoscopy (EGD), and it does not require capital equipment as magnetic endoscopy does. Flower offers the identification and location of bleeding sources in the stomach.

SUMMARY:
Clinical Study Overview Feasibility Study Plan (Study 1: Healthy Participants) Study 1- Confirming Flower capsule performance characteristics in detection of retained gastric contents greater than 1.5mL/kg in Healthy volunteers

1. Study Purpose

a. A controlled, prospective, between-participants study design to assess Flower in detecting the presence or absence of retained gastric contents (RGC), using sedated esophagogastroduodenoscopy (EGD) as the ground truth for an empty stomach and known ingested volume as the ground truth for a fed participant.

2. Study Endpoints

a. Primary i. Visualization of Retained Gastric Contents b. Secondary i. Gastric mucosal visualization of the seven anatomical landmarks of the stomach (fundus, cardia, lesser gastric curvature, greater gastric curvature, angulus, antrum, and pylorus) ii. Gastric Cleanliness iii. Adverse events defined as capsule retention, capsule aspiration, perforation, nausea, and pain iv. Maximum, tolerated water consumed v. Patient tolerance vi. Exploratory attempts for successful swallowing vii. Exploratory minimum and maximum water volume for optimal Flower performance viii. Time required for gastric examination completion by Flower

DETAILED DESCRIPTION:
There is an unmet clinical need for a rapid, accurate, and cost-effective tool to assess gastric content preoperatively, especially in high-risk populations such as individuals with obesity, diabetes, and those taking GLP-1 receptor agonists. The preoperative identification of retained gastric contents (RGC) is crucial in guiding anesthetic management, including the decision to perform endotracheal intubation, and in reducing the risk of aspiration-related complications.

The Flower System is a novel, single-use, wireless capsule endoscopy platform developed to provide real-time gastric imaging at the bedside without the need for sedation or advanced endoscopic infrastructure. The system consists of three key components: (1) the ingestible Flower capsule with an integrated high-resolution camera and software for orientational bias; (2) a wireless Dongle that receives and transmits video data to the physician's computer or smartphone; and (3) a software application with a user interface for image visualization, storage, and interpretation.

This clinical feasibility study evaluates the diagnostic performance and safety of the Flower capsule in two populations: (1) healthy volunteers (Study I), and (2) patients receiving GLP-1 receptor agonists (Study II; not described here). This protocol pertains to Study I only.

Study Design Overview - Study I This is a prospective, controlled, between-participant study comparing the diagnostic capability of the Flower capsule with sedated esophagogastroduodenoscopy (EGD), which serves as the ground truth standard for the presence or absence of gastric contents.

Twenty-four (n=24) healthy volunteers will be randomly assigned to one of two arms:

Group 1 - Empty Stomach Validation: Participants fast for 8 hours from solids and 2 hours from liquids, undergo sedated EGD to confirm an empty stomach, and then undergo Flower capsule evaluation.

Group 2 - Gastric Content Detection: Participants fast identically, undergo EGD to confirm an empty stomach, consume 1.5 mL/kg of a standardized semi-solid meal (post-alertness), and subsequently undergo Flower capsule evaluation.

A gastroenterologist blinded to fasting/fed status will assess the Flower capsule images for RGC and other endpoints.

Study Objectives Primary Objective: To determine the sensitivity and specificity of the Flower capsule in detecting RGC (>1.5 mL/kg) compared to the known ingested volume (fed group) and EGD (fasted group).

Secondary Objectives: To evaluate visualization of gastric landmarks, gastric cleanliness, safety (adverse events including capsule retention, aspiration, nausea, pain), water tolerance, examination duration, and patient-reported tolerance compared to EGD.

Technical Protocol All participants receive a structured hydration protocol using simethicone to minimize bubbles and improve mucosal visualization. Body position adjustments (supine, right lateral, left lateral, and prone) are used to achieve panoramic gastric visualization. The Flower capsule is orientationally biased to face upward, facilitating gravity-assisted mucosal inspection.

Participants are monitored for adverse events including capsule retention, aspiration, or signs of obstruction. Capsule passage is confirmed by participant-reported expulsion (with photographic evidence incentivized) and mandatory X-ray follow-up at 2 weeks post-procedure. In cases of non-expulsion, endoscopic or surgical retrieval will be arranged.

Evaluation Metrics Retained Gastric Contents: Binary detection (present/absent) based on image review.

Gastric Landmarks Visualized: Seven regions (fundus, cardia, lesser and greater curvatures, angulus, antrum, pylorus).

Mucosal Visualization Quality (4-point scale):

Grade 1: <50% Grade 2: ≥50% Grade 3: ≥75% Grade 4: ≥90%

Gastric Cleanliness Score (4-point scale):

Grade 1: Large debris/turbidity, no visualization Grade 2: Significant interference Grade 3: Minor interference Grade 4: Clear view Patient Tolerance Score (1-10): Lower scores indicate better experience. Adverse Events: Documented from Day 0 to follow-up (Day 14). Capsule Swallow Attempts and Total Exam Time: Tracked as feasibility markers. Follow-Up and Safety Monitoring

Participants are discharged same-day if stable. Safety surveillance includes:

Night-of follow-up call Daily calls from Day 1 to Day 7 for symptom checks Mandatory Day 14 follow-up with physical exam, vital signs, adverse event reporting, and abdominal X-ray Lost-to-follow-up is defined after three failed phone contact attempts and one certified letter to the last known address. All study-related procedures and follow-up visits are provided at no cost to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years and < 65 years (male or female)
2. Willing and able to sign an IEC-approved informed consent form
3. Willing and able to comply with all study requirements

Exclusion Criteria:

1. History of gastrointestinal disorders
2. History of gastroparesis
3. History of prior gastric surgery
4. Swallowing disorders
5. Contraindications to EGD or capsule endoscopy
6. Use of GLP-1 receptor agonists in the last 3 months
7. Diagnosed with diabetes mellitus
8. Classified as obese (based on BMI criteria)
9. Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-08 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Detection of Retained Gastric Contents Using Flower Capsule | Within 1 hour post-capsule ingestion
  Proportion of participants in whom the presence or absence of retained gastric contents (>1.5 mL/kg) is accurately identified using the Flower Capsule, compared to the reference standard (sedated EGD or known ingested volume).

SECONDARY OUTCOMES:
Visualization of Gastric Anatomical Landmarks | Within 1 hour post-capsule ingestion
  Number of gastric landmarks (fundus, cardia, lesser curvature, greater curvature, angulus, antrum, pylorus) successfully visualized using the Flower capsule.
Gastric Mucosal Visualization Score | Within 1 hour post-capsule ingestion
  Quality of mucosal visualization at each landmark based on a 4-point scale (1 = Poor, 4 = Excellent).
Gastric Cleanliness Score | Within 1 hour post-capsule ingestion
  Degree of gastric cleanliness based on a 4-point scale (1 = Poor, 4 = Excellent).
Adverse Events Related to Flower Capsule | From Day 0 to Day 14
  Number of participants with any of the following adverse events: capsule retention, aspiration, nausea, pain, perforation.
Time to Complete Gastric Examination | Within 1 hour post-capsule ingestion
  Total time required to complete Flower capsule-based gastric examination.
Capsule Swallowing Success | Within 15 minutes of capsule administration
  Number of attempts required to successfully swallow the Flower capsule.
Total Water Volume Consumed | Prior to capsule ingestion
  Total volume of water consumed to achieve adequate gastric distention prior to Flower examination.
Patient Tolerance Score for Flower Capsule | Immediately after Flower capsule examination
  Participant-reported tolerance using a 10-point scale (1 = best experience, 10 = worst experience).

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khandekar SS, Doctor JR, Awaskar SK, Alex NK, Medha LR, Ranganathan P. Ultrasound-guided estimation of gastric residual volume using Perlas's formula: A validation study in patients. Indian J Anaesth. 2022 Apr;66(4):255-259. doi: 10.4103/ija.ija_783_21. Epub 2022 Apr 20. PMID 35663207
- [Background] Silveira SQ, da Silva LM, de Campos Vieira Abib A, de Moura DTH, de Moura EGH, Santos LB, Ho AM, Nersessian RSF, Lima FLM, Silva MV, Mizubuti GB. Relationship between perioperative semaglutide use and residual gastric content: A retrospective analysis of patients undergoing elective upper endoscopy. J Clin Anesth. 2023 Aug;87:111091. doi: 10.1016/j.jclinane.2023.111091. Epub 2023 Mar 2. PMID 36870274
- [Background] Heckmann ND, Palmer R, Mayfield CK, Gucev G, Lieberman JR, Hong K. Glucagon-Like Peptide Receptor-1 Agonists Used for Medically-Supervised Weight Loss in Patients With Hip and Knee Osteoarthritis: Critical Considerations for the Arthroplasty Surgeon. Arthroplast Today. 2024 Jun 27;27:101327. doi: 10.1016/j.artd.2024.101327. eCollection 2024 Jun. PMID 39071832
- [Background] Chaitra TS, Palta S, Saroa R, Jindal S, Jain A. Assessment of residual gastric volume using point-of-care ultrasonography in adult patients who underwent elective surgery. Ultrasound J. 2023 Feb 8;15(1):7. doi: 10.1186/s13089-023-00307-8. PMID 36752856
- [Background] Warner MA, Meyerhoff KL, Warner ME, Posner KL, Stephens L, Domino KB. Pulmonary Aspiration of Gastric Contents: A Closed Claims Analysis. Anesthesiology. 2021 Aug 1;135(2):284-291. doi: 10.1097/ALN.0000000000003831. PMID 34019629
- [Background] Sharma G, Jacob R, Mahankali S, Ravindra MN. Preoperative assessment of gastric contents and volume using bedside ultrasound in adult patients: A prospective, observational, correlation study. Indian J Anaesth. 2018 Oct;62(10):753-758. doi: 10.4103/ija.IJA_147_18. PMID 30443057
- [Background] Son YG, Shin J, Ryu HG. Pneumonitis and pneumonia after aspiration. J Dent Anesth Pain Med. 2017 Mar;17(1):1-12. doi: 10.17245/jdapm.2017.17.1.1. Epub 2017 Mar 27. PMID 28879323